CLINICAL TRIAL: NCT02357017
Title: Mechanisms of Refractory Hypertension (High and Low Salt Diet)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in priority of interventional protocols
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Calhoun, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B000502641
Record Dates: First submitted 2015-01-22; First posted 2015-02-06 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low salt diet (Active Comparator): The low-salt meals will be formulated to provide 50 mmol of sodium per day. Two diets with different caloric amounts (2000 or 2500) will be available.
  Interventions: Dietary Supplement: NaCl tablets
- High salt diet (Active Comparator): High dietary salt intake, NaCl tablets (6 grams/day) will added to the subject's study diet in order to increase dietary sodium intake to >250 mmol/day.
  Interventions: Dietary Supplement: NaCl tablets

INTERVENTIONS:
Dietary Supplement: NaCl tablets

SUMMARY:
The purpose of the study is to test the hypothesis that persistent fluid retention and high sympathetic output contributes to the development of refractory hypertension (HTN). The investigators will determine, in a cross-over assessment of high and low salt diets, if dietary sodium restriction reduces 24-hr ambulatory BP in patients with refractory HTN. Moreover, the investigators will determine if dietary sodium restriction lessens the severity of obstructive sleep apnea (OSA) in patients with refractory HTN.

DETAILED DESCRIPTION:
We are proposing a unique phenotype of antihypertensive treatment failure that we refer to as refractory HTN. We have come to feel that while resistant (RHTN) represents a broad phenotype with multiple and overlapping etiologies of treatment resistance, there is a unique subset of patients who never achieve BP control in spite of maximal therapy. In a recently published retrospective analysis of our clinic experience, we found that patients with refractory HTN comprised about 10% of patients referred to us for RHTN.

A large number of intervention studies have verified the benefit of dietary salt restriction to reduce BP. We made such an assessment in a prospective, randomized, cross-over comparison of high- and low salt diets in 12 patients with confirmed RHTN. The average reduction in BP going from high to the low salt diet was 23/10 mmHg in the clinic and 20/10 mmHg during 24-hr ambulatory BP monitoring. These dramatic results demonstrated that patients with RHTN are exquisitely salt-sensitive and highlight the degree of BP reduction that can be accomplished with meaningful salt restriction. However, we are proposing the novel hypothesis that refractory HTN is mechanistically unique from RHTN in that it is not secondary to recalcitrant fluid retention.

Determining an association between dietary salt restriction and severity of obstructive sleep apnea (OSA) would potentially help us to find new therapies guided towards achieving better control of BP in patients with refractory HTN. We will investigate the effect of dietary salt intake on severity of OSA vascular function in patients with refractory HTN by doing vascular studies (pulse wave analysis/velocity, calculating thoracic impedance)).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥ 19 years of age
* Refractory hypertension defined as office BP > 140/90 that is uncontrolled with at least 5 different classes of antihypertensive medications
* Self-reported adherence >80% with prescribed antihypertensive medications

Exclusion Criteria:

* Severe hypertension (office BP >160/100 mm Hg)
* History of congestive heart failure (ejection fraction of <40%)
* Chronic kidney disease (creatinine clearance <60 ml/min)
* History of cardiovascular disease (stroke, TIA, myocardial infarction, or revascularization procedure)
* White coat hypertension defined as office BP >140/90 mm Hg and ambulatory daytime BP <135/85 mm Hg
* Pregnant or nursing women

Ages: 19 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour ambulatory systolic blood pressure (BP). | baseline to 4 weeks
  The mean change in blood pressure for each group after receiving 4 weeks of either a low salt diet compared to High dietary salt intake. The low-salt meals will be formulated to provide 50 mmol of sodium per day. Two diets with different caloric amounts (2000 or 2500) will be available. High dietary salt intake, NaCl tablets (6 grams/day) will added to the subject's study diet in order to increase dietary sodium intake to >250 mmol/day.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Calhoun, MD, Principal Investigator — Cardiology Department - University of Alabama at Birmingham